CLINICAL TRIAL: NCT05042479
Title: Using of Virtual Reality to Relieve Procedural Pain in Pediatric Oncology.
Acronym: VIRTUOSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: For Ever Fabien (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC21_0008
Record Dates: First submitted 2021-08-25; First posted 2021-09-13 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Hematologic Malignancy; Hematologic Non Malignancy; Solid Tumor, Childhood; Child, Only
Keywords: Pediatric; Pediatric oncology; Pain; Virtual reality; Nurse
MeSH Terms: conditions — Hematologic Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard treatment then virtual reality then choice between the two (Experimental): Efficiency of VR will be evaluated for each patient across 3 potentially painful care-procedures :
  For the first treatment, the child will benefit usual distraction and pain prevention techniques.
  For the 2nd, the child will use a VR headset as well as pain prevention techniques (excluding oxygen-nitrous oxide mixtures). The child will choose the application he/she wishes to use according to his/her age and parental agreement.
  For the 3rd treatment, the child will choose his/her favorite technique.
  Interventions: Other: Usual distraction and pain prevention techniques.; Other: Virtual reality; Other: Choice between usual distraction or virtual reality

INTERVENTIONS:
Other: Usual distraction and pain prevention techniques. — For the first painful procedure, the child will benefit usual distraction and pain prevention techniques.Pain prevention and management techniques commonly used in the conduct of care:
  * Application of a patch or anaesthetic cream 1 hour before the treatment
  * Vigilant sedation using a premedication for lumbar punctures: Midazolam /Nalbuphine/Hydroxyzine/Morphine.
  * Apart from care using VR, MEOPA can be given to the child for all assessed care on prescription.
  * Apart from care using VR, the usual distraction techniques are left to the patient's choice (electronic tablet, smartphone, games, songs...)
  * The presence of the parents
Other: Virtual reality — For the 2nd painful procedure, the child will use a VR (virtual reality) headset as well as pain prevention techniques (excluding oxygen-nitrous oxide mixtures). The child will choose the application he/she wishes to use according to his/her age.
Other: Choice between usual distraction or virtual reality — For the 3rd painful procedure, the child will choose his/her favorite technique between :
  Usual distraction and pain prevention techniques or virtual reality

SUMMARY:
Medical procedures can be a very frightening experience for children. It is known that children who received painful medical procedures can develop a higher sensitivity of pain during their following experiences.

During their treatments for malignant diseases, children are exposed to a lot of painful procedures (eg. needle insertion, lumbar punction, myelogram, etc…)

Therefore, medical societies propose the use of interventions like distraction techniques for pain management in complement of pharmacological treatment.

In addition, the repetitions of painful procedures and ineffective prevention of pain can create care phobia.

Within this context, immersive and participative virtual reality (VR) could be an innovative distraction technique for pain management among children undergoing medical procedures.

Attention Pain Theory can explain how virtual reality can reduce the perception of pain. Attention is required to feel pain. When the patient is focused on another subject like an immersive virtual environment, his brain is less available to treat information like painful stimulus from care procedures.

The investigators hypothesis is that VR can reduce procedural-related pain and can decrease fear during the following procedures.

Results of previous studies are varied : some showed a non-significant reduction of patient's procedural pain despite the use of VR, whereas others concluded to a decrease of pain. The question of the benefit of VR for the patients who are exposed to repeated painful procedures remains still unclear, especially with patients who are likely to feel chronic pain or many pain-related exposures.

The aim of this study is to evaluate the non-inferiority of virtual reality as a distraction technique for pain management in children and adolescents with onco-hematological diseases, undergoing painful procedures, compared to standard of care.

DETAILED DESCRIPTION:
VIRTUOSO is a study that aims to evaluate the impact of using a virtual reality headset to prevent care-induced pain in pediatric oncology. This study plans to include 34 patients. It is a single-center, non-inferiority, controlled, with cross-over study.

Efficiency of VR will be evaluated for each patient across 3 potentially painful care-procedures :

For the first treatment, the child will benefit usual distraction and pain prevention techniques.

For the 2nd treatment, the child will use a VR headset as well as pain prevention techniques (excluding oxygen-nitrous oxide mixtures). The child will choose the application he/she wishes to use according to his/her age.

For the 3rd treatment, the child will choose his/her favorite technique.

The virtual reality headset is an Occulus Quest headset, composed of 2 integrated earphones. It is adapted to the environment and can be used sitting or standing.

Usual pharmacological techniques for pain prevention will be maintained as per local practice.

All concomitant treatments are authorized except the use of oxygen-nitrous oxide mixtures.

The duration of this study is approximately 20 months. Inclusion will be for 10 months, patient follow-up for 6 months. Data analysis will be performed during 4 months.

During each treatment, if the child wishes to stop VR, the helmet will be removed and the usual techniques will be offered.

After each procedure, a self-assessment of the pain will be done immediately, using VAS.

At the end of the third treatment, a short questionnaire will be proposed to the child in order to collect the reasons for his choice. Another questionnaire will also be proposed to the parent present during the care.

A qualitative component will explore the social representations of the parents. A range of semi-directive interviews will be conducted with 6 families by a trained professional under the supervision of the methodologist.

ELIGIBILITY:
Inclusion Criteria:

Quantitative component:

* Child aged 7 to 18 years
* Child followed in pediatric onco-hematology in the context of hematological malignancy or non malignant hematology or solid tumor management.
* Child who has already experienced a potentially painful care procedure before entry the study
* Child who will have the same potentially painful care procedure (Hüber needle placement or lumbar puncture) on three occasions during the course of their care.
* Child with consent.
* Child whose parental authority holders have given their consent to participate to the study.

Qualitative component:

* Professional who used both care-induced pain prevention techniques and agreed to be interviewed.
* A parent or guardian.

Exclusion Criteria:

* Child who refuse to use this distraction technique (VR).
* Child who refuse to not use MEOPA during VR.
* Child who hasn't experienced the potentially painful care procedure that will be done during the study at least once before inclusion
* Child who does not speak French and whose parents do not speak French

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Pain level measured by VAS (self-evaluation) during the first care using standard treatment. | Immediately after the first care.
  Pain levels measured on the VAS. VAS : Visual Analogue Scale . Minimum value : 0. Maximum value : 10. The maximum value is the worse outcome.
Pain level measured by VAS (self-evaluation) during the second care using virtual reality | Immediately after the second care .
  Pain levels measured on the VAS. VAS : Visual Analogue Scale . Minimum value : 0. Maximum value : 10. The maximum value is the worse outcome.
Pain level measured by VAS (self-evaluation) during the third care using virtual reality or standard treatment | Immediately after the third care .
  Pain levels measured on the VAS. VAS : Visual Analogue Scale . Minimum value : 0. Maximum value : 10. The maximum value is the worse outcome.

SECONDARY OUTCOMES:
Percentage of children who choose VR in the 3rd care | Immediately after the 3rd intervention.
  Patient preference between VR and usual pain prevention technique for the same care.
  The difference between the pain level measured on a VAS with the use of VR and the pain level with the usual technique.
  VAS : Visual Analogue Scale . Minimum value : 0. Maximum value : 10. The maximum value is the worse outcome.
Patient questionnaire | Immediately after the 3rd intervention.
  Analysis of the answers to the patient questionnaire after treatment n°3. Description of the reasons for selecting the preferred technique.
Side effects to the use of VR | During each intervention with virtual reality (care 2 and care 3 if VR is chosen). Up to 6 months.
  Record of side effects reported in the e-CRF. Description of the potential side effects to the use of VR in care.
Ethnographic approach to caregivers' experiences after using the VR headset. | Through study completion - up to 20 months.
  Direct observation of the care unit. Understand the obstacles and levers for professionals to implement a new pain prevention device during care.
parent questionnaire. | Immediately after the 3rd intervention.
  Analysis of the responses to the parent questionnaire. Understand parents' experience of care when implementing a new pain prevention device during care.
Thematic analysis of the verbatim collected during the semi-directive interviews with the parents after Care 3 | Immediately after the 3rd intervention.
  Understand the social representations of parents and children regarding the use of a virtual reality device.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes CHU, Nantes, France